CLINICAL TRIAL: NCT05299892
Title: Optimizing Soft Speech Recognition in Children With Hearing Loss
Acronym: SoftSpeech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Hearts for Hearing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 458
Record Dates: First submitted 2022-03-01; First posted 2022-03-29 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Intervention Model Description: One group of participants will be assessed unaided and aided with Phonak Audeo P or Phonak Naida P hearing aids with Speech Enhancer "off", "on at moderate", and "on at strong" settings.
Masking Description: Participants will be "blind" as to whether the Speech Enhancer feature is activated or deactivated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Children with Hearing Loss (Experimental): Participants age 5-12 with hearing loss who will be fit with study hearing aids and tested on speech perception in unaided and aided condition.
  Interventions: Device: Phonak Audeo P or Naida P hearing aid

INTERVENTIONS:
Device: Phonak Audeo P or Naida P hearing aid — Commercially available hearing aid that has access to speech enhancer feature settings "off", "moderate" and "strong"

SUMMARY:
Overhearing is important for vocabulary learning and speech and language development in young children. However, contemporary hearing aids are generally unable to provide adequate access to low-level auditory inputs from multiple talkers at a distance to capitalize on overhearing. A recent investigation by Jace Wolfe and colleagues showed that, even when aided, children with hearing loss had significantly poorer speech recognition at 40, 50 and 60 dBA compared to children with normal hearing. Furthermore, they showed that increasing hearing aid gain for very low-level inputs produced a statistically significant improvement in syllable-final plural recognition and a non-significant trend toward better monosyllabic word recognition at very low presentation levels. Additional research is needed to document low-level speech recognition ability of children with hearing loss as well as the potential benefit or detriment of increasing hearing aid gain for low-level inputs. A novel hearing aid technology known as Soft Speech Enhancer has been shown improve low-level speech perception in adults with hearing loss; however, the effect of Speech Enhancer on speech recognition in children is not yet known and will be evaluated.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate whether soft speech recognition in quiet is significantly improved with Speech Enhancer (SE) "on" at the default setting (moderate) compared to Speech Enhancer "off" in children with moderate (N3) to severe (N5) hearing loss. There are several secondary objectives: 1) To evaluate the main effects of age and Speech Enhancer strength, and potential interaction on speech recognition and comfort in children with moderate to severe hearing loss. 2) To demonstrate that hearing aids compensate for hearing loss in children.

This confirmatory clinical investigation will be executed at Hearts for Hearing. It is a single-group, single blind intervention study with each participant serving as his or her own control. However, in certain conditions participant blinding is not feasible (i.e., aided versus unaided performance). The outcome measures being assessed include: speech recognition in quiet with Consonant-Nucleus-Consonant (CNC) words, and comfort ratings using a Multiple Stimuli with Hidden Reference and Anchor (MUSHRA) procedure and looped sentences overlaid with low-level transient noise.

Four different hearing aid conditions will be assessed in this clinical investigation: unaided (no amplification), aided with SE "off", aided with SE "moderate", aided with SE "strong". For the unaided or no treatment condition no hearing aids will be worn. For aided conditions, experienced hearing aid users will be fit binaurally with investigational devices matching their personal device form factor connected to their personal acoustic coupling (e.g., earmold). Using the Audioscan Verifit 2, probe microphone measurements will be conducted to match DSL 5.0 pediatric quiet and noise targets. Three distinct programs will be created, each with a different SE strength.

Hearing aid program order (speech enhancer settings) will be randomized for all testing conditions except for CNC at 50 dBA Quiet with SE Off; that condition is administered first to establish candidacy for further testing. A randomized list of SE settings was generated for all participants for the remaining conditions.

Testing will be completed in a double-walled sound booth with calibrated equipment. Recorded stimuli will be presented through loudspeakers (Sony CFD-ZW755) from clinical audiometers (Grayson Stadler Standard) or Dell computers using the Arizona State University Speech Recognition Program, Windows Media Player and Adobe Audition. Speech stimuli will be presented from a loudspeaker located at 0 degrees azimuth (directly in front).

Speech recognition results will be compared to determine the effect of amplification on accuracy scores as well as the influence of speech enhancer on behaviorally measured benefit and subjectively-derived listening preference.

ELIGIBILITY:
Inclusion Criteria:

* native English speakers who communicate verbally
* no known speech language disorders, cognitive or learning issues
* experienced hearing aid users (> 6 months use)
* "full-time" hearing aid users (i.e., wear on a daily basis)
* CNC word scores of 30% or better at 50dBA in quiet with SE "off"

Exclusion Criteria:

* new hearing aid users
* inconsistent hearing aid users
* <4 years or >12 years of age
* non-native English speaker who communicates verbally
* known cognitive/ learning issues or speech language disorder
* CNC word scores < 30% correct presented at 50dBA in quiet with SE "off"

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hearts for Hearing, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hearing Impaired Users: Hearing impaired children, age 5 -12 years who are fit with either Audeo P or Naida P and complete all testing requirements (unaided, aided with SE off, aided with SE on moderate, and aided with SE on strong).
Period: Overall Study
Arm/Group | Hearing Impaired Users
Started | 36
Completed | 34
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Participants who were enrolled in study and were fit with the study hearing aids.
Groups:
- Children With Hearing Loss, Age 5-12: Participants age 5-12 with hearing loss who will be fit with study hearing aids and tested on speech perception in all four required conditions: Unaided, Aided with SE off, Aided with SE moderate, and Aided with SE strong.
  Phonak Audeo P or Naida P hearing aid: Commercially available hearing aid that has access to speech enhancer feature settings "off", "moderate" and "strong"
Arm/Group | Children With Hearing Loss, Age 5-12
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 9 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Speech Recognition in Quiet Using CNC (Consonant-Nucleus-Consonant) Word Lists
Description: One word list of 25 words is presented at 50 dB (quiet conditions) through a front speaker. The percent correctly repeated words are calculated and a higher score indicates better speech perception. The participants completed this task without hearing aids. Data was collected on both age groups, but analysis was completed only on the entire group as a whole. Age effects were not tested.
Time Frame: Day 1 of 1 day study
Population: Hearing impaired participants who completed all required testing conditions: 1) word recognition unaided, 2)word recognition at 40 dB input with SE off, 3) word recognition at 40 dB input with SE on moderate setting, 4) word recognition at 40 dB input with SE on strong setting, 5) word recognition at 50 dB input with SE off, 6) word recognition with at 50 dB input with SE on moderate setting, and 7) word recognition with 50 dB input with SE on strong setting.
Measure: Mean (Standard Deviation); unit: percentage of correctly repeated words
Groups:
- Hearing Impaired Children Age 5-12: Hearing impaired children, age 5 -12 years who are fit with either Audeo P or Naida P and tested in all four required conditions: unaided condition at 50 dB, and aided condition with SE off, on at moderate, and on at strong at 40 and 50 dB.
Arm/Group | Hearing Impaired Children Age 5-12
Number analyzed (Participants) | 33
percentage of correctly repeated words
  Percent words correct unaided, in quiet (50 dBA) | 6.06 (9.73)
  Percent words correct aided with SE off, in quiet ( 40 dBA) | 53.7 (13.02)
  Percent words correct, aided with SE moderate, in quiet (40 dBA) | 66.61 (11.92)
  Percent words correct, aided with SE strong, in quiet (40 dBA) | 69.7 (12)
  Percent words correct, aided SE off, in quiet (50 dBA) | 74.7 (9.1)
  Percent words correct, aided SE moderate, in quiet (50 dBA) | 81.76 (6.78)
  Percent words correct, aided SE strong, in quiet (50 dBA) | 83.76 (6.87)
Statistical Analysis 1: Comparison: Hearing Impaired Children Age 5-12; An ANOVA was conducted for the three SE conditions (off, moderate, strong) at 50 dBA .Post -hoc comparisons were done using Bonferroni's correction. Below result is the mean comparison between SE of and SE moderate. Analysis of age effects was not completed; Test type: Other; p = .005, ANOVA; Mean Difference (Final Values) = 6.46153, 95% CI 2-sided [1.79 to 12.99]
Statistical Analysis 2: Comparison: Hearing Impaired Children Age 5-12; An ANOVA was conducted for the three SE conditions (off, moderate, strong) at 50 dBA . Post -hoc comparisons were done using Bonferroni's correction. Below result is the mean comparison between SE of and SE strong. An analysis of age effects was not completed; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 9.00961, 95% CI 2-sided [3.91 to 15.11]
Statistical Analysis 3: Comparison: Hearing Impaired Children Age 5-12; Null hypothesis: There will be no significant differences between the mean unaided CNC score at 50 dBA and the mean aided CNC score with SE off; Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Subjective Ratings of Speech Enhancer
Description: Participants will listen to a sound sample of looped sentences overlaid with low-level transient noise with the Speech Enhancer at different settings (off, moderate, strong) and rate their preference. An A/B comparison will be used to compare Speech Enhancer Off vs. Speech Enhancer Moderate, and Speech Enhancer Off vs. Speech Enhancer Strong. Participants answered three questions: 1) Which sounds better?, 2) Which is more comfortable?, and 3) Which do you prefer? Results will be reported as qualitative data and no statistical analysis will take place.
Time Frame: Day 1 of 1 day study
Population: All participants who completed the testing requirements and were able to provide answers to all three questions: 1) Which sounds better? 2) Which is more comfortable? and 3) Which do you prefer? Data was collected on both age groups, but was analysis was completed only on entire group as a whole. Age effects were not analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Hearing Impaired Users Age 5 -12: Hearing impaired children, age 5 -12 years who are fit with either Audeo P or Naida P and tested in all required conditions: unaided condition, and aided condition with SE off, on at moderate, and on at strong and were able to answer all three questions.
Arm/Group | Hearing Impaired Users Age 5 -12
Number analyzed (Participants) | 32
Participants
  SE Moderate sounds better than SE Off | 10
  SE Moderate sounds the same as SE Off | 16
  SE Off sounds better than SE Moderate | 6
  SE Moderate is more comfortable than SE Off | 6
  SE Moderate is the same comfort as SE Off | 14
  SE Off is more comfortable than SE Moderate | 12
  Prefer SE Moderate to SE Off | 12
  Prefer both SE Off and SE Moderate the same | 12
  Prefer SE Off to SE Moderate | 8
  SE Strong sounds better than SE Off: number analyzed (Participants) | 31
  SE Strong sounds better than SE Off | 15
  SE Strong sounds the same as SE Off: number analyzed (Participants) | 31
  SE Strong sounds the same as SE Off | 11
  SE Off sounds better than SE Strong: number analyzed (Participants) | 31
  SE Off sounds better than SE Strong | 5
  SE Strong is more comfortable than SE Off: number analyzed (Participants) | 31
  SE Strong is more comfortable than SE Off | 8
  SE Strong is the same comfort as SE Off: number analyzed (Participants) | 31
  SE Strong is the same comfort as SE Off | 17
  SE Off is more comfortable than SE Strong: number analyzed (Participants) | 31
  SE Off is more comfortable than SE Strong | 6
  Prefer SE Strong to SE Off: number analyzed (Participants) | 31
  Prefer SE Strong to SE Off | 16
  Prefer both SE Strong and SE Off the same: number analyzed (Participants) | 31
  Prefer both SE Strong and SE Off the same | 9
  Prefer SE Off to SE Strong: number analyzed (Participants) | 31
  Prefer SE Off to SE Strong | 6

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Children With Hearing Loss
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT05299892/Prot_SAP_001.pdf